CLINICAL TRIAL: NCT00814580
Title: A Randomized, Double-Blind, Multi-Center, Parallel-Group Study of Tapentadol Immediate Release (IR) Versus Oxycodone IR for the Treatment of Subjects With Acute Post-Operative Pain Following Elective Arthroscopic Shoulder Surgery
Brief Title: Safety and Efficacy of Tapentadol Immediate Release (IR) and Oxycodone IR for Treatment of Acute Post-op Pain Following Elective Arthroscopic (Surgery Using a Thin Flexible Scope) Shoulder Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015040; R331333PAI3022 (Other: Ortho-McNeil Janssen Scientific Affairs, LLC); KF5503/49 (Other: Grunenthal GmbH)
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Results first posted 2012-01-10 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Postoperative Pain
Keywords: analgesia; postoperative pain; opioid; rotator cuff repair; labral tear repair; Bankart procedure; oxycodone; tapentadol; arthroscopic shoulder surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Tapentadol IR First dose: one 50 mg capsule (a re-dose of 50 mg is permitted as soon as one hour after the first dose on Day 1 if needed) Subsequent doses: one or two capsules (50 mg or 100 mg) every 4 to 6 hours as needed
  Interventions: Drug: Tapentadol IR
- 002 (Active Comparator): Oxycodone IR First dose: one 5 mg capsule (a re-dose of 5 mg is permitted as soon as one hour after the first dose on Day 1 if needed Subsequent doses: one or two capsules (5 mg or 10 mg) every 4 to 6 hours as needed
  Interventions: Drug: Oxycodone IR

INTERVENTIONS:
Drug: Tapentadol IR — First dose: one 50 mg capsule (a re-dose of 50 mg is permitted as soon as one hour after the first dose on Day 1, if needed) Subsequent doses: one or two capsules (50 mg or 100 mg) every 4 to 6 hours as needed
  Arms: 001
Drug: Oxycodone IR — First dose: one 5 mg capsule (a re-dose of 5 mg is permitted as soon as one hour after the first dose on Day 1, if needed Subsequent doses: one or two capsules (5 mg or 10 mg) every 4 to 6 hours as needed
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate how tapentadol immediate release (IR) and oxycodone IR treat moderate to severe post-operative pain after elective arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
This is a double-blind (neither the patient nor the study doctor knows the name of the assigned study drug during the study), randomized (study drug selected by chance like flipping a coin), active-comparator (patient will get active drug and there is no inactive drug), outpatient study to evaluate efficacy and how well a patient tolerates multiple doses of tapentadol immediate release (IR) versus oxycodone IR for short-term moderate to severe post-operative pain after arthroscopic (a surgical technique whereby a doctor inserts a tube-like instrument into a joint to visually inspect and repair tissues) shoulder surgery. About 370 patients will be enrolled to either receive tapentadol IR or oxycodone IR until approximately 150 patients in each treatment group are enrolled. After obtaining informed consent, patients will have screening visit procedures to determine study eligibility. Visit 1 (screening) may begin up to 21 days prior to surgery. Pre-operative assessments (e.g., physical examinations, clinical laboratory assessments) will be conducted as part of routine procedures. Patients will have a urine drug test and women who are able to have children will have a urine pregnancy test performed as part of screening prior to the study. Height and weight will be taken and a sleep questionnaire will also be completed at screening. Study staff will conduct pre-operative teaching regarding post-operative pain including: the pain intensity assessment for the study (11-point numeric rating scale where 0=no pain and 10=pain as bad as you can imagine); descriptions of mild, moderate and severe pain; instructions for dosing with study medication; and completing the study diary. Eligible patients will be post-operative men and women who have undergone elective outpatient arthroscopic shoulder surgery. Patients must have received a regional interscalene (within the scalene muscles) nerve block as the primary anesthetic (numbing medication) during the procedure and do not require intravenous (through a vein) patient-controlled analgesia post-operatively. Patients who are expected to have moderate to severe acute post-operative pain from shoulder surgery and who are appropriate candidates for outpatient pain management with an oral opioid (narcotic) pain medication will be eligible. In addition, appropriate patients are expected to require oral opioid pain medication post-operatively. Patients who continue to meet all study criteria post-operatively will be assigned to a study drug group prior to PACU discharge (PACU is considered Visit 2) and will be sent home with study medication. All patients will be prescribed a standard regimen of cold pack application to the surgical shoulder. Patients will be instructed to take the first dose of study medication as their first oral pain medication when they have at least "moderate" pain (prior to discharge or at home). Patients will be reminded about instructions on post-operative pain that were discussed during the pre-operative screening visit. Patients will also be instructed to complete a diary assessment of their current pain intensity before taking the first dose of study medication. Day 1 will be the calendar day when the patient takes the first dose of study medication. Starting on Day 1, patients will be instructed to complete assessments in paper diaries each morning and evening related to pain intensity, pain relief, and occurrences of vomiting. All patients will be contacted by telephone by a member of the study staff on the day following surgery. The staff will verify that the first dose of study medication was taken and the baseline pain intensity assessment was recorded. All patients will receive a second telephone call from the study staff on Day 3. During this telephone call, site personnel will inquire about the patient's overall status and will reinforce diary compliance. If the study staff determines it is necessary, the patient will be required to return to the study site for an unscheduled visit. Patients may take up to 2 pills (any form) of acetaminophen for pain other than post-operative shoulder pain (e.g., headache, back pain) once per day only for up to a total of 2 days during the study. Patients who take up to 325 mg/day aspirin as prevention for a heart condition will be permitted to enter the study and continue on study medication provided they are on a stable dose for at least 1 month prior to study entry and plan to continue the same dose during the study. Patients who complete the study will return to the study site for a final visit (Visit 3) on Day 7. Patients who discontinue early for any reason (i.e., lack of efficacy, adverse events, patient's choice) should contact the study staff before taking supplemental pain medication and schedule his/her final visit. Patients will complete a final assessment of pain intensity and pain relief. In addition, all patients will complete a sleep questionnaire, a Patient Global Impression of Change and an assessment of satisfaction with treatment. The study doctor will complete a Clinician Global Impression of Change and will record any medical resource utilization noted in the office charts (e.g., unplanned calls from the subject, unscheduled office visits, emergency room visits). Vital signs will be obtained and study medication will be collected and counted. Patients will have adverse events assessed and any changes in concomitant medications (other medications taken at the same time as the study medication) recorded. All patients will have post-study medication prescribed at the study doctor's discretion. A patient may elect to take supplemental pain medication to treat their post-operative shoulder pain at any time during the study; however, patients who take supplemental pain medication will be considered discontinued from the study. Patients will be assigned by chance equally (1:1) in a blinded (neither the patient or study doctor knows) fashion to get tapentadol immediate release (IR) 50 or 100 mg vs oxycodone IR 5 or 10 mg, every 4-6 hours as needed. Treatment is up to 7 days starting on Day 1 with one capsule of study medication. A "re-dose" is permitted and may be administered as soon as one hour after the first dose only. For subsequent doses, patients may take one or two capsules every 4 to 6 hours as needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and vital signs and meeting the American Society of Anesthesiology (ASA) physical status I, II, or III
* completed screening procedures and have undergone one of the following elective outpatient arthroscopic surgical procedures: rotator cuff repair, labral tear repair, Bankart repair
* an arthroscopic mini-open rotator cuff repair
* (an arthroscopic distal clavicle resection performed in conjunction with a rotator cuff, labral tear or Bankart repair is also permitted)
* received anesthesia administered to the shoulder by interscalene nerve block
* receive study medication as the first oral analgesic medication following the orthopedic surgical procedure and expected to have moderate to severe pain requiring oral opioids for at least 3 days after surgery.

Exclusion Criteria:

* Patients whose post-operative pain would require non opioid analgesia as standard of care
* received a non-allowed procedure
* received intraoperative or post-operative anesthesia and/or analgesic medications which are expected to provide post-operative analgesia for >24 hours after discharge from the PACU (recovery room)
* received intraoperatively >200 mg fentanyl or the morphine equivalent of another opioid (for the total procedure) or potent inhaled anesthesia (e.g., sevoflurane, isoflurane)
* received IV PCA analgesia (intravenous pump the patient controls) in the PACU or a PACU stay >8 hours
* expected to require inpatient treatment in a hospital or rehabilitation unit post operatively
* anticipate any surgical procedure(s) within 7 days after the initial shoulder surgery
* have significant nausea and/or vomiting at the time of randomization (patients may receive an anti-emetic prior to or during surgery)
* received any of the following: long-acting or controlled-release opioids within 1-month prior to randomization
* immediate release CII opioid formulations (e.g., Opana IR, Percocet, Percodan, oxycodone IR, Dilaudid) for >5 days total within 1 month before, and within 24 hours of, randomization
* intra-articular (within a joint) or systemic steroids (except inhalers and topical steroids), within 1 month before randomization (exception, patients on a stable dose of chronic steroids for a minimum of 3 months, for a condition other than the shoulder pain)
* use of non-steroidal anti-inflammatory drugs (NSAIDs) within 24-hours of randomization
* have taken any CIII opioid formulation (e.g., Tylenol with Codeine) >3 days/week in the 1-month prior to randomization
* treated with anticonvulsants, monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), neuroleptics, or serotonin norepinephrine reuptake inhibitors (SNRIs) within 2 weeks before randomization
* positive urine drug screen (cocaine, methadone, amphetamines, cannabinoids, opiates, benzodiazepines, barbiturates, and oxycodone)
* have an active systemic or local infection
* significant co-existing autoimmune inflammatory conditions
* history of seizure disorder or epilepsy
* presence of any of the following: mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of screening
* severe traumatic brain injury, episode(s) of unconsciousness of more than 24 hours duration, or post-traumatic amnesia of more than 24 hours duration within 15 years of screening
* known history of alcohol or drug abuse in the study doctor's judgment based on medical history
* known or suspected to be opioid tolerant or dependent
* known history of laboratory values reflecting severe kidney disease, known history of moderately or severely impaired liver function
* history of allergy to, or hypersensitivity to tapentadol, oxycodone, or other components of the medication
* history (within the past 6 months) of a major psychiatric disorder
* history of suicidal ideation or suicidal attempts within the past 2 years
* currently involved in litigation regarding their shoulder injury, have a disability claim or patients who are receiving Worker's Compensation due to their shoulder injury or are being evaluated to receive disability or Worker's Compensation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC

REFERENCES:
- [Derived] Vorsanger GJ, Klopfer AM, Xiang J, Benson CJ, Moskovitz BL, Rosenthal NR. Immediate-release tapentadol or oxycodone for treatment of acute postoperative pain after elective arthroscopic shoulder surgery: a randomized, phase IIIb study. J Opioid Manag. 2013 Jul-Aug;9(4):281-90. doi: 10.5055/jom.2013.0170. PMID 24353022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this outpatient, multicenter US only study occurred between Jan. 14, 2009 and Mar. 19, 2010
Pre-assignment Details: The study consisted of a screening period (up to 21 days) and a double-blind active treatment period (7 days, but can be up to 9 days).
Groups:
- Tapentadol IR: Tapentadol IR 50 or 100 mg 4-6 hours as needed; maximum 600mg a day for 7 days but can be up 9 days
- Oxycodone IR: Oxycodone IR 5 or 10 mg 4-6 hours as needed, maximum 60 mg a day for 7 days but can be up to 9 days
Period: Overall Study
Arm/Group | Tapentadol IR | Oxycodone IR
Started | 194 | 188
Completed | 163 | 141
Not Completed | 31 | 47
Not completed — Adverse Event | 6 | 15
Not completed — Lack of Efficacy | 18 | 25
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Other | 1 | 3
Not completed — Did Not Take Drug | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol IR | Oxycodone IR | Total
Number analyzed (Participants) | 192 | 186 | 378
Age, Categorical [Count of Participants; unit: Participants] — The summary statistics provided for baseline characteristic was based on safety population that includes 192 subjects in tapentadol group and 186 subjects in oxycodone group. The safety population includes randomized subjects took at least one dose of study drug.
  Participants
    <=18 years | 4 | 6 | 10
    Between 18 and 65 years | 138 | 137 | 275
    >=65 years | 50 | 43 | 93
Age Continuous [Mean (Standard Deviation); unit: years] — The summary statistics provided for baseline characteristic was based on safety population that includes 192 subjects in tapentadol group and 186 subjects in oxycodone group. The safety population includes randomized subjects took at least one dose of study drug.
  years | 53.2 (14.98) | 52.7 (14.97) | 52.9 (14.96)
Sex: Female, Male [Count of Participants; unit: Participants] — The summary statistics provided for baseline characteristic was based on safety population that includes 192 subjects in tapentadol group and 186 subjects in oxycodone group. The safety population includes randomized subjects took at least one dose of study drug.
  Participants
    Female | 69 | 58 | 127
    Male | 123 | 128 | 251
Region of Enrollment [Number; unit: participants] — The summary statistics provided for baseline characteristic was based on safety population that includes 192 subjects in tapentadol group and 186 subjects in oxycodone group. The safety population includes randomized subjects took at least one dose of study drug.
  participants
    USA | 192 | 186 | 378

OUTCOME MEASURES:

1. Primary Outcome: Summary and Analysis of Sum of Pain Intensity Difference (SPID) (With Imputation) Over 3 Days (72 Hours)
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID72 was calculated as the time-weighted Sum of PID scores over 72 hours. The range of SPID72 is from -720 to 720. The higher value in SPID indicates greater pain relief.
Time Frame: 3 Days (72 hours)
Population: The modified Intent-to-Treat(mITT) population was defined as all randomized subjects who took at least one dose of study drug within 24 hours of randomization and had a baseline pain intensity score >= 4 on an 11-point numeric rating scale (NRS).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 34.8 (134.18) | 40.5 (155.41)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Tapentadol IR versus Oxycodone IR; Test type: Non-Inferiority or Equivalence — Primary hypothesis test for non-inferiority of tapentadol IR over oxycodone IR required that upper limit of 95% CI for LS mean difference (oxycodone IR minus tapentadol IR) was less than the inferiority margin (< 72). If the upper limit was less than 0 then tapentadol IR was superior to oxycodone IR for SPID over 3 days at a 5% level of significance; p = 0.5265, ANCOVA — Analysis of covariance (ANCOVA) model included baseline pain intensity score as the covariate and treatment and pooled center as class variables; Least square mean difference = 9.0, 95% CI 2-sided [-18.9 to 36.9], Standard Error of Mean 14.2

2. Secondary Outcome: Summary of Kaplan-Meier Estimates for Time to Achieve 50% Reduction in Pain Intensity From Baseline
Description: From date of first administration of study medication to time to achieve adequate 50% reduction in pain intensity from baseline score. Censored observations included subjects who completed or discontinued from the study without a 50% reduction in pain intensity from baseline score. If a subject discontinued due to lack of efficacy (including rescue medication), the subject was censored on Day 7, 12 PM.
Time Frame: 7 Days
Population: Modified Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Hours | 125.3 [100.3 to NA] — NA: Not Applicable, as not enough participants achieved 50% pain reduction and upper limit of confidence interval. | NA [99.9 to NA] — NA: Not Applicable, as not enough participants achieved 50% pain reduction and upper limit of confidence interval.
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.7306, Log Rank

3. Secondary Outcome: Summary of Kaplan-Meier Estimates for Time to Achieve 30% Reduction in Pain Intensity From Baseline
Description: From date of first administration of study medication to time to achieve adequate 30% reduction in pain intensity from baseline score. Censored observations included subjects who completed or discontinued from the study without a 30% reduction in pain intensity from baseline score. If a subject discontinued due to lack of efficacy (including rescue medication), the subject was censored on Day 7, 12 PM.
Time Frame: 7 Days
Population: Modified Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Hours | 73.9 [54.5 to 89.0] | 66.4 [46.0 to 134.2]
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.8524, Log Rank

4. Secondary Outcome: Summary of 30% Responder Rate (With Imputation) on Day 3
Description: The 30% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 30% from baseline in pain intensity at Day 3 (average of Day 3 PM and Day 4 AM). If a subject has only the Day 3 PM value or Day 4 AM value, then response rate will be based on the non-missing value. If a subject withdraws or uses rescue medication before Day 3 PM then Baseline Observation Carried Forward (BOCF) will be imputed. Last Observation Carried Forward (LOCF) may be used if no value afterward.
Time Frame: Day 3
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
percentage of participants | 33.5 | 34.4
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.9078, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test (Row Mean Score option) controlling for pooled investigator centers

5. Secondary Outcome: Summary of 30% Responder Rate (With Imputation) on Day 7
Description: The 30% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 30% from baseline in pain intensity at Day 7 (average of Day 6 PM and Day 7 AM). If a subject has only the Day 6 PM value or Day 7 AM value, then response rate will be based on the non-missing value. If a subject withdraws or uses rescue medication before Day 6 PM then BOCF will be imputed. LOCF may be used if no value afterward.
Time Frame: Day 7
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
percentage of participants | 48.1 | 42.2
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.2633, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test (Row Mean Score option) controlling for pooled investigator centers

6. Secondary Outcome: Summary of 50% Responder Rate (With Imputation) on Day 3
Description: The 50% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 50% from baseline in pain intensity at Day 3 (average of Day 3 PM and Day 4 AM). If a subject has only the Day 3 PM value or Day 4 AM value, then response rate will be based on the non-missing value. If a subject withdraws or uses rescue medication before Day 3 PM then BOCF will be imputed. LOCF may be used if no value afterward.
Time Frame: Day 3
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
percentage of participants | 19.0 | 22.7
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.4498, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test (Row Mean Score option) controlling for pooled investigator centers

7. Secondary Outcome: Summary of 50% Responder Rate (With Imputation) on Day 7
Description: The 50% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 50% from baseline in pain intensity at Day 7 (average of Day 6 PM and Day 7 AM). If a subject has only the Day 6 PM value or Day 7 AM value, then response rate will be based on the non-missing value. If a subject withdraws or uses rescue medication before Day 6 PM then BOCF will be imputed. LOCF may be used if no value afterward.
Time Frame: Day 7
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
percentage of participants | 35.4 | 29.2
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.2158, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test (Row Mean Score option) controlling for pooled investigator centers

8. Secondary Outcome: Summary and Analysis of Sum of Pain Intensity Difference (SPID) (With Imputation) Over 2 Days (48 Hours)
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID48 was calculated as the time-weighted Sum of PID scores over 48 hours. The range of SPID48 is from -480 to 480. The higher value in SPID indicates greater pain relief.
Time Frame: 2 Days (48 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 10.6 (88.05) | 14.6 (102.24)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.4811, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = 6.6, 95% CI 2-sided [-11.8 to 25.0], Standard Error of Mean 9.34

9. Secondary Outcome: Summary and Analysis of Sum of Pain Intensity Difference (SPID) (With Imputation) Over 7 Days
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID over 7 Days was calculated as the time-weighted Sum of PID scores up to Day 7, 8 AM. The range is from -1440 to 1440. The higher value in SPID indicates greater pain relief.
Time Frame: 7 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 136.1 (277.20) | 122.1 (299.87)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.7405, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = -9.3, 95% CI 2-sided [-64.7 to 46.0], Standard Error of Mean 28.13

10. Secondary Outcome: Summary and Analysis of Total Pain Relief (TOTPAR) (With Imputation) Over 2 Days (48 Hours)
Description: Pain Relief was defined as a 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum over all pain relief up to hour 48. The range of TOTPAR over 2 days is from 0 to 192. A higher value in TOTPAR indicated greater pain relief.
Time Frame: 2 Days (48 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 97.7 (48.13) | 92.0 (50.74)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.3097, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = -5.6, 95% CI 2-sided [-16.5 to 5.3], Standard Error of Mean 5.53

11. Secondary Outcome: Summary and Analysis of Total Pain Relief (TOTPAR) (With Imputation) Over 3 Days (72hours)
Description: Pain Relief was defined as a 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum over all pain relief up to hour 72. The range of TOTPAR over 3 days is from 0 to 288. A higher value in TOTPAR indicated greater pain relief.
Time Frame: 3 Days (72hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 151.3 (71.9) | 140.9 (77.39)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.2179, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = -10.3, 95% CI 2-sided [-26.7 to 6.1], Standard Error of Mean 8.34

12. Secondary Outcome: Summary and Analysis of Total Pain Relief (TOTPAR) (With Imputation) Over 7 Days
Description: Pain Relief was defined as a 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum over all pain relief up to Day 7, 8 AM. The range of TOTPAR over 7 days is from 0 to 576. A higher value in TOTPAR indicated greater pain relief.
Time Frame: 7 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 299.1 (137.33) | 272.9 (154.31)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.1051, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = -26.3, 95% CI 2-sided [-58.1 to 5.5], Standard Error of Mean 16.16

13. Secondary Outcome: Summary and Analysis of the Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) (With Imputation) Over 2 Days (48 Hours)
Description: The Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) was derived from Sum of TOTPAR and SPID. The range of SPRID over 2 days is from -480 to 672. A higher value in SPRID indicated greater pain relief.
Time Frame: 2 Days (48 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 108.2 (109.89) | 106.6 (125.82)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.9367, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = 1.0, 95% CI 2-sided [-22.8 to 24.8], Standard Error of Mean 12.09

14. Secondary Outcome: Summary and Analysis of the Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) (With Imputation) Over 3 Days (72 Hours)
Description: The Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) was derived from Sum of TOTPAR and SPID. The range of SPRID over 3 days is from -720 to 1008. A higher value in SPRID indicated greater pain relief.
Time Frame: 3 Days (72hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 186.1 (168.64) | 181.4 (193.97)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.9441, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = -1.3, 95% CI 2-sided [-37.8 to 35.2], Standard Error of Mean 18.53

15. Secondary Outcome: Summary and Analysis of the Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) (With Imputation) Over 7 Days
Description: The Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) was derived from Sum of TOTPAR and SPID. The range of SPRID over 7 days is from -1440 to 2016. A higher value in SPRID indicated greater pain relief.
Time Frame: 7 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 158 | 154
Scores on a scale | 435.2 (354.59) | 395.0 (386.16)
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.3427, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least square mean difference = -35.6, 95% CI 2-sided [-109.3 to 38.1], Standard Error of Mean 37.45

16. Secondary Outcome: Subject Satisfaction With Treatment
Description: Treatment satisfaction was measured using a 7-point scale where 1 = very satisfied and 7 = very dissatisfied
Time Frame: 7 Days
Population: Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 192 | 181
percentage of participants
  Very satisfied | 58.3 | 48.1
  Somewhat satisfied | 15.6 | 20.4
  Slightly satisfied | 2.6 | 5.5
  Neither satisfied nor dissatisfied | 7.3 | 5.0
  Slightly dissatisfied | 3.6 | 3.3
  Somewhat dissatisfied | 2.1 | 1.7
  Very dissatisfied | 9.9 | 14.4
  Missing | 0.5 | 1.7
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.1618, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test (row mean score option) controlling for pooled investigator centers

17. Secondary Outcome: Patient Global Impression of Change (PGIC) at End of Study
Description: Patient Global Impression of Change (PGIC) was defined as the 7-point numeric scale, where 1=very much improved to 7=very much worse.
Time Frame: 7 Days
Population: Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 192 | 181
percentage of participants
  Very much improved | 27.6 | 26.0
  Much improved | 46.9 | 42.5
  Minimally improved | 15.6 | 13.3
  No change | 3.1 | 7.7
  Minimally worse | 2.1 | 2.2
  Much worse | 1.6 | 0.6
  Very much worse | 1.0 | 5.5
  Missing | 2.1 | 2.2
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.0481, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test (row mean score option) controlling for pooled investigator centers

18. Secondary Outcome: Clinician Global Impression of Change (CGIC) at End of Study
Description: Clinician Global Impression of Change (CGIC) was defined as the 7-point numeric scale, where 1=very much improved to 7=very much worse.
Time Frame: 7 Days
Population: Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 192 | 181
percentage of participants
  Very much improved | 33.3 | 29.3
  Much improved | 47.4 | 39.8
  Minimally improved | 11.5 | 12.7
  No change | 3.6 | 7.2
  Minimally worse | 1.0 | 2.2
  Much worse | 1.0 | 1.1
  Very much worse | 1.0 | 5.0
  Missing | 1.0 | 2.8
Statistical Analysis 1: Comparison: Tapentadol IR vs Oxycodone IR; Test type: Superiority or Other; p = 0.0109, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test (row mean score option) controlling for pooled investigator centers

19. Secondary Outcome: Summary of Medical Resource Utilization - Number of Calls by the Subject to Study Site Personnel
Description: Information associated with contacts with a healthcare professional was collected by the investigator and study staff for all subjects throughout the study.
Time Frame: 7 Days
Population: Intent-to-Treat Population
Measure: Number; unit: Number of calls
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 192 | 181
Number of calls
  Total number of subjects who made calls | 69 | 74
  Number of adverse event related calls | 39 | 28
  Number of pain-related calls | 46 | 70
  Number of non-medical/administrative calls | 16 | 19
  Number of other medical conditions calls | 10 | 7
  Total number of calls | 105 | 122

20. Secondary Outcome: Summary of Medical Resource Utilization - Number of Other Types of Contacts With Healthcare Professionals
Description: as for outcome 19
Time Frame: 7 Days
Population: Intent-to-Treat Population
Measure: Number; unit: Number of participants
Arm/Group | Tapentadol IR | Oxycodone IR
Number analyzed (Participants) | 192 | 181
Number of participants
  Patients visited a healthcare professional | 87 | 89
  Number of patient with scheduled visits | 84 | 85
  Number of patient with unscheduled visits | 7 | 6
  Number of patient with Internist | 2 | 1
  Number of patient with Orthopedic surgeon | 80 | 87
  Number of patient with Physical therapist | 3 | 0
  Number of patient with Primary care physician | 5 | 1
  Patient with other healthcare professional | 2 | 1
  Number of patient with emergency room visit | 6 | 6
  Number of patient with hospital admissions | 0 | 2

21. Secondary Outcome: Sleep Quality: Trouble Falling Asleep? - Shift of Measurement From Baseline to End of Study (Tapentadol IR)
Description: Over the past 7 days patients reported "trouble falling asleep" by using a 4-category scale (not at all, 1 to 2 days, 3 to 5 days, 6 to 7 days) at baseline and the final study visit (Day 7).
Time Frame: Baseline and 7 Days
Population: Tapentadol IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Groups:
- End of Study: Not at All: Tapentadol IR participants who chose category of 'Not at all' for the measurement at the end of study.
- End of Study: 1-2 Days: Tapentadol IR participants who chose category of '1-2 Days' for the measurement at the end of study.
- End of Study: 3-5 Days: Tapentadol IR participants who chose category of '3-5 Days' for the measurement at the end of study.
- End of Study: 6-7 Days: Tapentadol IR participants who chose category of '6-7 Days' for the measurement at the end of study.
- Baseline - Total: Total Tapentadol IR participants at the baseline.
- End of Study: Missing the Measurement: Tapentadol IR Participants who missed the measurement at the end of study.
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 63 | 56 | 35 | 35 | 192 | 3
participants
  Baseline: Not at all | 34 | 34 | 20 | 16 | 104 | 0
  Baseline: 1-2 Days | 15 | 12 | 7 | 5 | 40 | 1
  Baseline: 3-5 Days | 8 | 6 | 4 | 6 | 26 | 2
  Baseline: 6-7 Days | 5 | 4 | 4 | 8 | 21 | 0
  Baseline: Miss the measurement | 1 | 0 | 0 | 0 | 1 | 0

22. Secondary Outcome: Sleep Quality: Trouble Falling Asleep? - Shift of Measurement From Baseline to End of Study (Oxycodone IR)
Description: as for outcome 21
Time Frame: Baseline and 7 Days
Population: Oxycodone IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Groups:
- End of Study: Not at All: Oxycodone IR participants who chose category of 'Not at all' for the measurement at the end of study.
- End of Study: 1-2 Days: Oxycodone IR participants who chose category of '1-2 Days' for the measurement at the end of study.
- End of Study: 3-5 Days: Oxycodone IR participants who chose category of '3-5 Days' for the measurement at the end of study.
- End of Study: 6-7 Days: Oxycodone IR participants who chose category of '6-7 Days' for the measurement at the end of study.
- Baseline - Total: Total Oxycodone IR participants at the baseline.
- End of Study: Missing the Measurement: Oxycodone IR Participants who missed the measurement at the end of study.
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 67 | 45 | 33 | 32 | 181 | 4
participants
  Baseline: Not at all | 44 | 23 | 21 | 14 | 105 | 3
  Baseline: 1-2 Days | 11 | 12 | 4 | 7 | 34 | 0
  Baseline: 3-5 Days | 7 | 8 | 3 | 5 | 24 | 1
  Baseline: 6-7 Days | 3 | 2 | 5 | 6 | 16 | 0
  Baseline: Miss the measurement | 2 | 0 | 0 | 0 | 2 | 0

23. Secondary Outcome: Sleep Quality: Wake up Several Times During Night? - Shift of Measurement From Baseline to End of Study (Tapentadol IR)
Description: Over the past 7 days patients reported "Wake up several times during night" by using a 4-category scale (not at all, 1 to 2 days, 3 to 5 days, 6 to 7 days) at baseline and the final study visit (Day 7).
Time Frame: Baseline and 7 Days
Population: Tapentadol IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 20 | 48 | 42 | 79 | 192 | 3
participants
  Baseline: Not at all | 9 | 12 | 8 | 12 | 42 | 1
  Baseline: 1-2 Days | 2 | 12 | 8 | 13 | 35 | 0
  Baseline: 3-5 Days | 3 | 17 | 12 | 21 | 53 | 0
  Baseline: 6-7 Days | 5 | 7 | 14 | 33 | 61 | 2
  Baseline: Miss the measurement | 1 | 0 | 0 | 0 | 1 | 0

24. Secondary Outcome: Sleep Quality: Wake up Several Times During Night? - Shift of Measurement From Baseline to End of Study (Oxycodone IR)
Description: as for outcome 23
Time Frame: Baseline and 7 Days
Population: Oxycodone IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 17 | 36 | 45 | 79 | 181 | 4
participants
  Baseline: Not at all | 8 | 14 | 6 | 14 | 44 | 2
  Baseline: 1-2 Days | 5 | 7 | 11 | 23 | 46 | 0
  Baseline: 3-5 Days | 2 | 11 | 10 | 12 | 36 | 1
  Baseline: 6-7 Days | 2 | 3 | 18 | 29 | 53 | 1
  Baseline: Miss the measurement | 0 | 1 | 0 | 1 | 2 | 0

25. Secondary Outcome: Sleep Quality: Trouble Staying Asleep? - Shift of Measurement From Baseline to End of Study (Tapentadol IR)
Description: Over the past 7 days patients reported "Trouble staying asleep" by using a 4-category scale (not at all, 1 to 2 days, 3 to 5 days, 6 to 7 days) at baseline and the final study visit (Day 7).
Time Frame: Baseline and 7 Days
Population: Tapentadol IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 50 | 47 | 45 | 47 | 192 | 3
participants
  Baseline: Not at all | 27 | 24 | 17 | 13 | 81 | 0
  Baseline: 1-2 Days | 12 | 13 | 7 | 8 | 41 | 1
  Baseline: 3-5 Days | 5 | 3 | 13 | 9 | 31 | 1
  Baseline: 6-7 Days | 5 | 7 | 8 | 17 | 38 | 1
  Baseline: Miss the measurement | 1 | 0 | 0 | 0 | 1 | 0

26. Secondary Outcome: Sleep Quality: Trouble Staying Asleep? - Shift of Measurement From Baseline to End of Study (Oxycodone IR)
Description: as for outcome 25
Time Frame: Baseline and 7 Days
Population: Oxycodone IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 46 | 40 | 34 | 57 | 181 | 4
participants
  Baseline: Not at all | 26 | 17 | 12 | 20 | 77 | 2
  Baseline: 1-2 Days | 8 | 13 | 8 | 13 | 42 | 0
  Baseline: 3-5 Days | 5 | 6 | 7 | 9 | 29 | 2
  Baseline: 6-7 Days | 6 | 3 | 7 | 14 | 30 | 0
  Baseline: Miss the measurement | 1 | 1 | 0 | 1 | 3 | 0

27. Secondary Outcome: Sleep Quality: Pain Interferes With Sleep? - Shift of Measurement From Baseline to End of Study (Tapentadol IR)
Description: Over the past 7 days patients reported "Pain interferes with sleep" by using a 4-category scale (not at all, 1 to 2 days, 3 to 5 days, 6 to 7 days) at baseline and the final study visit (Day 7).
Time Frame: Baseline and 7 Days
Population: Tapentadol IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 50 | 59 | 46 | 34 | 192 | 3
participants
  Baseline: Not at all | 23 | 17 | 13 | 2 | 56 | 1
  Baseline: 1-2 Days | 13 | 17 | 9 | 5 | 46 | 2
  Baseline: 3-5 Days | 6 | 15 | 10 | 7 | 38 | 0
  Baseline: 6-7 Days | 7 | 10 | 14 | 20 | 51 | 0
  Baseline: Miss the measurement | 1 | 0 | 0 | 0 | 1 | 0

28. Secondary Outcome: Sleep Quality: Pain Interferes With Sleep? - Shift of Measurement From Baseline to End of Study (Oxycodone IR)
Description: as for outcome 27
Time Frame: Baseline and 7 Days
Population: Oxycodone IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 27 | 52 | 50 | 48 | 181 | 4
participants
  Baseline: Not at all | 16 | 15 | 15 | 9 | 57 | 2
  Baseline: 1-2 Days | 4 | 11 | 15 | 6 | 37 | 1
  Baseline: 3-5 Days | 3 | 16 | 6 | 5 | 31 | 1
  Baseline: 6-7 Days | 4 | 8 | 14 | 28 | 54 | 0
  Baseline: Miss the measurement | 0 | 2 | 0 | 0 | 2 | 0

29. Secondary Outcome: Sleep Quality: Wake up Feeling Tired and Worn Out? - Shift of Measurement From Baseline to End of Study (Tapentadol IR)
Description: Over the past 7 days patients reported "Wake up feeling tired and worn out" by using a 4-category scale (not at all, 1 to 2 days, 3 to 5 days, 6 to 7 days) at baseline and the final study visit (Day 7).
Time Frame: Baseline and 7 Days
Population: Tapentadol IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 53 | 51 | 47 | 38 | 192 | 3
participants
  Baseline: Not at all | 35 | 19 | 8 | 9 | 71 | 0
  Baseline: 1-2 Days | 8 | 16 | 17 | 6 | 49 | 2
  Baseline: 3-5 Days | 4 | 10 | 14 | 8 | 36 | 0
  Baseline: 6-7 Days | 5 | 6 | 8 | 15 | 35 | 1
  Baseline: Miss the measurement | 1 | 0 | 0 | 0 | 1 | 0

30. Secondary Outcome: Sleep Quality: Wake up Feeling Tired and Worn Out? - Shift of Measurement From Baseline to End of Study (Oxycodone IR)
Description: as for outcome 29
Time Frame: Baseline and 7 Days
Population: Oxycodone IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 51 | 46 | 44 | 36 | 181 | 4
participants
  Baseline: Not at all | 28 | 23 | 20 | 8 | 82 | 3
  Baseline: 1-2 Days | 14 | 12 | 13 | 9 | 48 | 0
  Baseline: 3-5 Days | 3 | 8 | 6 | 6 | 24 | 1
  Baseline: 6-7 Days | 4 | 3 | 5 | 13 | 25 | 0
  Baseline: Miss the measurement | 2 | 0 | 0 | 0 | 2 | 0

31. Secondary Outcome: Sleep Quality: Feeling Alert During Daytime Hours? - Shift of Measurement From Baseline to End of Study (Tapentadol IR)
Description: Over the past 7 days patients reported "Feeling alert during daytime hours" by using a 4-category scale (not at all, 1 to 2 days, 3 to 5 days, 6 to 7 days) at baseline and the final study visit (Day 7).
Time Frame: Baseline and 7 Days
Population: Tapentadol IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 16 | 41 | 63 | 69 | 192 | 3
participants
  Baseline: Not at all | 3 | 6 | 3 | 11 | 23 | 0
  Baseline: 1-2 Days | 1 | 6 | 8 | 9 | 24 | 0
  Baseline: 3-5 Days | 7 | 10 | 14 | 10 | 41 | 0
  Baseline: 6-7 Days | 5 | 19 | 38 | 38 | 103 | 3
  Baseline: Miss the measurement | 0 | 0 | 0 | 1 | 1 | 0

32. Secondary Outcome: Sleep Quality: Feeling Alert During Daytime Hours? - Shift of Measurement From Baseline to End of Study (Oxycodone IR)
Description: as for outcome 31
Time Frame: Baseline and 7 Days
Population: Oxycodone IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 24 | 31 | 51 | 71 | 181 | 4
participants
  Baseline: Not at all | 5 | 3 | 4 | 12 | 25 | 1
  Baseline: 1-2 Days | 2 | 5 | 9 | 3 | 20 | 1
  Baseline: 3-5 Days | 3 | 6 | 13 | 12 | 34 | 0
  Baseline: 6-7 Days | 14 | 17 | 25 | 42 | 100 | 2
  Baseline: Miss the measurement | 0 | 0 | 0 | 2 | 2 | 0

33. Secondary Outcome: Sleep Quality: Feeling Well Rested? - Shift of Measurement From Baseline to End of Study (Tapentadol IR)
Description: Over the past 7 days patients reported "Feeling well rested" by using a 4-category scale (not at all, 1 to 2 days, 3 to 5 days, 6 to 7 days) at baseline and the final study visit (Day 7).
Time Frame: Baseline and 7 Days
Population: Tapentadol IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 36 | 35 | 59 | 59 | 192 | 3
participants
  Baseline: Not at all | 11 | 7 | 9 | 11 | 39 | 1
  Baseline: 1-2 Days | 9 | 9 | 9 | 7 | 34 | 0
  Baseline: 3-5 Days | 7 | 13 | 20 | 14 | 55 | 1
  Baseline: 6-7 Days | 9 | 6 | 21 | 26 | 63 | 1
  Baseline: Miss the measurement | 0 | 0 | 0 | 1 | 1 | 0

34. Secondary Outcome: Sleep Quality: Feeling Well Rested? - Shift of Measurement From Baseline to End of Study (Oxycodone IR)
Description: as for outcome 33
Time Frame: Baseline and 7 Days
Population: Oxycodone IR arm of Intent-to-Treat population. Shift table from baseline to end of study (Day 7).
Measure: Number; unit: participants
Arm/Group | End of Study: Not at All | End of Study: 1-2 Days | End of Study: 3-5 Days | End of Study: 6-7 Days | Baseline - Total | End of Study: Missing the Measurement
Number analyzed (Participants) | 34 | 44 | 45 | 54 | 181 | 4
participants
  Baseline: Not at all | 10 | 6 | 4 | 6 | 27 | 1
  Baseline: 1-2 Days | 4 | 11 | 11 | 5 | 32 | 1
  Baseline: 3-5 Days | 9 | 14 | 14 | 13 | 50 | 0
  Baseline: 6-7 Days | 11 | 13 | 15 | 29 | 70 | 2
  Baseline: Miss the measurement | 0 | 0 | 1 | 1 | 2 | 0

ADVERSE EVENTS:
Arm/Group | Tapentadol IR | Oxycodone IR
Serious Adverse Events (participants affected / at risk) | 0/192 | 3/186
Other Adverse Events (participants affected / at risk) | 83/192 | 75/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol IR (N=192) | Oxycodone IR (N=186)
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol IR (N=192) | Oxycodone IR (N=186)
Vomiting (Gastrointestinal disorders) | 36 | 19
Nausea (Gastrointestinal disorders) | 33 | 30
Constipation (Gastrointestinal disorders) | 17 | 27
Headache (Nervous system disorders) | 18 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 15

LIMITATIONS AND CAVEATS:
No notable study limitations were identified by the Sponsor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days